CLINICAL TRIAL: NCT04250844
Title: Use of Intrapyloric Botulinum Injections in Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Rachel Rosen, Associate Professor of Pediatrics, Boston Children's Hospital
Other Study IDs: P00033019
Record Dates: First submitted 2020-01-23; First posted 2020-01-31 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Vomiting; Feeding Disorders; Gastroparesis
Keywords: Botulinum Toxin
MeSH Terms: conditions — Vomiting; Feeding and Eating Disorders; Gastroparesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Botulinum: We will follow for symptom improvement over time patients with nausea, vomiting, feeding intolerance, or other signs of gastric dysfunction who were determined by their gastroenterologist to require upper endoscopy with intrapyloric botulinum injections and if clinically applicable endoscopic functional luminal imaging probe (EndoFLIP). The dosage will be determined by the patient's physician.
- Control: We will follow for symptom improvement over time patients with nausea, vomiting, feeding intolerance, or other signs of gastric dysfunction who were determined by their gastroenterologist to require upper endoscopy without intrapyloric botulinum injections.

SUMMARY:
This study aims to evaluate the effect of intrapyloric botulinum toxin in children with feeding disorders.

DETAILED DESCRIPTION:
Chronic vomiting and feeding difficulties are common in young children and have a negative physical and psychosocial impact for patients and families. Currently there is no straightforward treatment algorithm for these issues, and management often involves multiple medication trials and procedures. Intrapyloric botulinum toxin injection has been proposed as a treatment for nausea and vomiting in adults, but there is minimal prior research on use in children and no prior research on use in children with feeding disorders. The aims of this study are: (1) to determine the efficacy of intrapyloric botulinum toxin injection for reducing gastrointestinal symptoms in children, (2) to determine the efficacy of intrapyloric botulinum injections for improving feeding outcomes in children, and (3) to define predictors of response to intrapyloric botulinum toxin injection.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic nausea, vomiting, or feeding intolerance undergoing upper endoscopy with or without intrapyloric botulinum injections.
* Age between 30 days and 18 years.

Exclusion Criteria:

* Significant uncontrolled inflammation on upper or lower endoscopy
* Known inflammatory bowel disease
* Uncontrolled thyroid disease
* Current opioid use

Ages: 30 Days to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients from our tertiary care center who are undergoing upper endoscopy with or without intrapyloric botulinum injections.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-03-10 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Degree of improvement in quality of life | 4 weeks
  Quality of life will be measured with the Pediatric Quality of Life Inventory (PedsQL). This is composed of 23 items comprising 4 dimensions: Physical Functioning, Emotional Functioning, Social Functioning, and School Functioning. Each item is answered using a 3-point scale: 0 (Not at all), 2 (Sometimes), 4 (A lot). Scores range 0 to 100, with lower scores indicating worse quality of life. The outcome will be assessed by calculating the change in score from baseline to 4 weeks.

SECONDARY OUTCOMES:
Degree of symptomatic improvement | 4 weeks
  Symptoms will be measured with the Gastroparesis Cardinal Symptom Index (GCSI). The GCSI is based on three subscales: post-prandial fullness/early satiety (4 items); nausea/vomiting (3 items), and bloating (2 items). A six-point Likert response scale, ranging from 0 (none) to 5 (very severe) is used to rate severity of each symptom. Scores range from 0 to 45, with higher scores indicating worse symptoms. This outcome will be assess by calculating the change in score from baseline to 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Rosen, MD, MPH, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No